CLINICAL TRIAL: NCT06464653
Title: The Efficacy and Safety of Pallidothalamic Tracts Electrical Stimulation for Lennox-Gastaut Syndrome: A Prospective, Pilot Trial
Brief Title: Pallidothalamic Tracts Electrical Stimulation for Lennox-Gastaut Syndrome
Acronym: PESL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liankun_Ren (Other)
Responsible Party: Sponsor-Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-128-003
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-12

CONDITIONS: Lennox Gastaut Syndrome
Keywords: Deep Brain Stimulation; Lennox-Gastaut Syndrome; Pallidothalamic Tracts
MeSH Terms: conditions — Lennox Gastaut Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pallidothalamic Tracts-DBS group (Experimental): participants will undergo Pallidothalamic Tracts-DBS ON with the individual stimulation parameters determined in the parameter determination period, then continue to receive stimulation for the remainder of the study.
  Interventions: Device: Forel's Field H-DBS ON

INTERVENTIONS:
Device: Forel's Field H-DBS ON — The surgical intervention named deep brain stimulation is a well-established neurosurgical treatment for drug-resistant epilepsy. The targets used in this study is Forel's Field H. The devices used for intervention have been approved by Chinese National Medical Products Administration (CFDA). The postoperative drug dosage adjustment depends on the efficacy of DBS and the judgment of the epilepsy specialist.

SUMMARY:
The primary objective of this research is to study the efficacy and safety of deep brain stimulation (DBS) of pallidothalamic tracts as adjunctive therapy for alleviating symptoms in Lennox-Gastaut Syndrome.

DETAILED DESCRIPTION:
This project aims to include 5 participants, and evaluate the effectiveness and safety of pallidothalamic tracts stimulation in patients with Lennox-Gastaut Syndrome through a prospective, interventional, unblinded, single-arm clinical trial. It is expected to provide new therapeutic options for patients with Lennox-Gastaut Syndrome with alternative treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for Lennox-Gastaut Syndrome (LGS) based on comprehensive assessment of medical history, seizure semiology, and electroencephalographic (EEG) findings during both ictal and interictal periods;
2. Interictal EEG demonstrates generalized paroxysmal fast activity (GPFA) and slow spike-and-wave (SSW) complexes;
3. Generalized tonic-clonic seizures (GTCs) have been captured in prior video-EEG monitoring, or seizure episodes have been clearly described by reliable eyewitnesses;
4. During the screening or baseline period, the following conditions are met:

   1. The patient or caregiver is capable of reliably maintaining a seizure diary;
   2. The seizure diary indicates an average of at least 5 seizures per month;
   3. The patient is on two or more antiepileptic drugs (AEDs), with a stable treatment regimen (no new add-on or withdrawal of AEDs, excluding temporary rescue medications such as benzodiazepines; dose adjustments are allowed);
5. The patient has been evaluated through a comprehensive presurgical epilepsy workup and is considered unsuitable for, or has declined, resective epilepsy surgery, or has had unsatisfactory outcomes from resective or ablative procedures;
6. Providation of written informed consent, demonstrates adequate compliance with the study protocol, and agrees to participate in this clinical study.

Exclusion Criteria:

1. Unable to provide a reliable seizure diary by self or legal guardian;
2. Predominant seizure type is focal impaired awareness seizures;
3. Psychogenic non-epileptic seizures within 12 months;
4. Brain structual abnormalities precluding safe implantation of deep brain stimulator;
5. Conditions associated with increased risk of intraoperative or postoperative bleeding (e.g., coagulopathy), or requirement for long-term oral anticoagulant or antiplatelet therapy;
6. Presence of other severe somatic or internal medical conditions, including significant hepatic or renal dysfunction;
7. Pregnant, or planning to pregnant within 2 years.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Seizure Frequency (SF28) | Up to 1 year after Forel's Field H-DBS
  Seizure frequency (SF28) is defined as seizure count per month (28-day) period. The SF28 is calculated as follows, where D=total number of days for which seizure information is collected for the specific 28-day interval:
  SF28=(Total number of seizures in D days/D)*28. In addition, the baseline seizure frequency is defined as mean of 3- month SF28 in the baseline period. The seizure frequency in double-blind phase is defined as SF28 per month during the double-blind period. Percent change in seizure frequency=100*(double-blind SF28-baseline SF28)/baseline SF28.

SECONDARY OUTCOMES:
Seizure Responder Rate | Up to 1 year after Forel's Field H-DBS
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Life quality evaluation | Up to 1 year after Forel's Field H-DBS
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score. The minimum and maximum values, and whether higher scores mean a better or worse outcome.
Cognitive function evaluation (MMSE) | Up to 1 year after Forel's Field H-DBS
  Percentage change from baseline in Mini-Mental State Examination (MMSE) score. The MMSE score ranges from 0 to 30, with higher scores representing better cognitive function and lower scores indicating greater cognitive impairment.
Cognitive function evaluation (MoCA) | Up to 1 year after Forel's Field H-DBS
  Percentage change from baseline in Montreal Cognitive Assessment (MoCA) score. The MoCA score ranges from 0 to 30, with higher scores indicating better cognitive function and lower scores suggesting greater cognitive impairment.
Adverse Events | Up to 1 year after Pallidothalamic Tracts-DBS
  Rate of adverse events which were judged to be study-related throughout the study.
Incidence of Sudden Unexpected Death in Epilepsy (SUDEP) | Up to 1 year after Forel's Field H-DBS
  The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No